CLINICAL TRIAL: NCT04454580
Title: Retrospective, Observational, Monocentric Study to Assess Efficacy and Safety of the Combination of an Hypomethylating Agent in Combination With Venetoclax for Newly Diagnosed Acute Myeloid Leukemia Patients Not Eligible for Intensive Chemotherapy
Brief Title: Hypomethylating Agents and Venetoclax in Newly Diagnosed Acute Myeloid Leukemia Patients Not Eligible for Intensive Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Maggiore Di Trieste (Other)
Responsible Party: Principal Investigator, Francesco Zaja, Professor, Ospedale Maggiore Di Trieste
Other Study IDs: HMA-V
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia, Adult; Hypomethylating Agents; Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Decitabine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treated patients: hypomethylating agent (azacitidine or decitabine) in combination with venetoclax
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — treatment with azacitidine or decitabine in combination with venetoclax
  Other Names: Azacitidine; Decitabine

SUMMARY:
This is a retrospective, observational, monocentric study to evaluate the efficacy and safety of the combination of an hypomethylating agent with venetoclax newly diagnosed patients with acute myeloid leukemia ineligible for intensive chemotherapy

DETAILED DESCRIPTION:
The prognosis of acute myeloid leukemia (AML) patients who are ineligible for intensive chemotherapy is poor (Kantarjian et al). Hypomethylating agents, azacitidine and decitabine, are effective and less toxic regimens, and treatment with these agents has improved the prognosis of these patients (Fenaux et al).

Venetoclax, a Bcl-2 inhibitor, in combination with azacitidine has shown efficacy in AML patients with complete remission rate of 73% and overall survival at 2 years of 40-50% (Di Nardo et al).

On these grounds, the aim of this study is to collect the real-life experience with this combination in previously untreated AML patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* newly diagnosed acute myeloid leukemia not eligible for intensive chemotherapy

Exclusion Criteria:

* promyelocytic acute myeloid leukemia
* patients who have already received one or more prior lines of therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients with newly diagnosed acute myeloid leukemia not eligible for intensive chemotherapy, treated in a referral center for hematology
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | every three months after started treatment up to two years
  according to European Leukemia Network (ELN)

SECONDARY OUTCOMES:
Overall response rate (ORR) | every three months after started treatment up to two years
  according to European Leukemia Network (ELN)
Morphologic leukemia-free state (MLFS) | every three months after started treatment up to two years
  according to European Leukemia Network (ELN)
Progression-free-survival | from the start of the treatment until the date of documented progression or date of death from any cause, assessed up to 2 years
  from start of the treatment to progression or death
Overall survival | from the start of the treatment until the date of documented progression or date of death from any cause, assessed up to 2 years
  from start of the treatment to progression or death
adverse events and serious adverse events | through study completion, for an average of 1 year
  according to CTCAE v. 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Professor, Principal Investigator — SC Ematologia Ospedale Maggiore Trieste
Locations (1):
- SC Ematologia Ospedale Maggiore, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Result] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Result] Kantarjian H, Ravandi F, O'Brien S, Cortes J, Faderl S, Garcia-Manero G, Jabbour E, Wierda W, Kadia T, Pierce S, Shan J, Keating M, Freireich EJ. Intensive chemotherapy does not benefit most older patients (age 70 years or older) with acute myeloid leukemia. Blood. 2010 Nov 25;116(22):4422-9. doi: 10.1182/blood-2010-03-276485. Epub 2010 Jul 28. PMID 20668231